CLINICAL TRIAL: NCT04938986
Title: Interest of the Immunoscore® as a Post-operative Complementary Tool for the Detection of the Risk of Recurrence in Patients With Nonmetastatic Colorectal Cancer : Prospective Cohort Comparing the Recommandation for Patient Care According to the Immunoscore® With the Standard Care Decision.
Brief Title: Interest of the Immunoscore® as a Post-operative Complementary Tool for the Detection of the Risk of Recurrence in Patients With Nonmetastatic Colorectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PPC-IS
Record Dates: First submitted 2021-06-22; First posted 2021-06-25 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Non Metastatic Colorectal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMMUNOSCORE® (Experimental)
  Interventions: Diagnostic Test: IMMUNOSCORE®

INTERVENTIONS:
Diagnostic Test: IMMUNOSCORE® — recommendation for patient care according to the result of the IMMUNOSCORE®

SUMMARY:
Evaluate the patient care recommandation induced by the IMMUNOSCORE® result

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 inclusive;
* histologically confirmed colon adenocarcinoma;
* having undergone a curative resection of stage I, II or III colorectal cancer;
* diagnosed T1 / T2 / T3 / T4 and N0 / N1 / N2;
* eligible to receive 6 months of adjuvant chemotherapy;
* having given free, informed and written consent;
* agreeing to the use of a tumor sample for research purposes;
* being affiliated to a social security system.

Exclusion Criteria:

* pregnant or breastfeeding women
* legal incapacity or physical, psychological, social or geographical conditions preventing the patient from signing the consent or completing the study.
* history of other solid tumor within 3 years before inclusion, with the exception of in-situ cancer of the cervix and skin cancers (basal or squamous) treated and controlled
* person subject to a safeguard measure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Number of cases where the recommendations for patient care according to the Immunoscore® are considered beneficial compared to the standard care decision | 5 years

SECONDARY OUTCOMES:
Replication error (RER) phenotype | 6 and 9 months
  Number of cases where the Immunoscore® resultat is inconsistent with the RER phenotype
KRAS, NRAS and BRAF mutations | 6 and 9 months
  Number of cases where the Immunoscore® resultat is inconsistent with the KRAS, NRAS and BRAF mutations
Ratio of ciruclating tumor DNA level | 6 and 9 months
  Number of cases where the Immunoscore® resultat is inconsistent with the ratio of ciruclating tumor DNA level
Actual survival (patient alive without recurrence, alive with recurrence, dead) | 5 years
  Number of cases where the Immunoscore® resultat is inconsistent with the actual survival

CONTACTS AND LOCATIONS:
Overall Officials: Hervé PERRIER, M.D, Principal Investigator — Hopital Saint Joseph Marseille; Yves RINALDI, M.D, Principal Investigator — Hopital Européen Marseille
Locations (2):
- France (2):
  - Hôpital Européen, Marseille
  - Hopital Saint Joseph, Marseille